CLINICAL TRIAL: NCT06620549
Title: Feasibility of Nurse-performed Gastric Point-of-care Ultrasound to Determine Gastric Content After Gastro-intestinal and Oncologic Surgery: a Pilot Study
Brief Title: Feasibility of Nurse-performed Gastric Ultrasound After Surgery
Acronym: SKILLS-2
Status: Recruiting | Type: Observational
Sponsor: Radboud University Medical Center (Other)
Responsible Party: Sponsor
Other Study IDs: 2024-17217
Record Dates: First submitted 2024-04-16; First posted 2024-10-01 (Actual); Last update posted 2024-10-01 (Actual); Status verified 2024-04

CONDITIONS: Point-of-care-ultrasound; Gastric Ultrasonography; Gastric Ultrasound; Gastro Intestinal Surgery; Nursing; Abdominal Surgeries

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Patients after gastro-intestinal surgery: Postoperative patients after gastro-intestinal surgery (e.g. liver, pancreatic, colorectal or hyperthermic intraperitoneal chemotherapy (HIPEC) surgery)
  Interventions: Diagnostic Test: gastric ultrasonograppy

INTERVENTIONS:
Diagnostic Test: gastric ultrasonograppy — Patients will be scanned in both supine and right lateral decubitus position (RLD)s. If the antrum is visible, it will be judged if the antrum is empty in both positions or the antrum is empty in supine position and fluid apparent in RLD position suggesting a low fluid volume (<1,5 ml/Kg). The third option is fluid apparent in both supine and RLD position, suggesting a higher fluid volume (>1,5ml/Kg) and the last option is solid food in one or both positions.

SUMMARY:
Gastric ultrasound is a quick and non-invasive tool to evaluate gastric content.

Emptying of gastric content can be affected after abdominal surgery leading to the inability of tolerating oral foods. Gastric content can be assessed by gastric ultrasound and nurses were recently trained to do so in healthy volunteers; however, feasibility of nurse-performed gastric ultrasound after major abdominal surgery is not investigated yet.

This study aims to investigate the feasibility of nurse-performed gastric point-of-care ultrasound after major gastro-intestinal surgery.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients (>18 years)
* Underwent gastrointestinal surgery:

  * partial liver resection,
  * colorectal resection,
  * HIPEC,
  * pancreatic procedures including Whipple procedures for pancreatic cancer or pancreatic disorders,
  * other gastro- intestinal abdominal procedures such as resections of sarcomas, correction of herniation.
* Obtained written informed consent.
* Admitted for at least 3 days.

Exclusion Criteria:

* patients with open abdominal wounds or with abdominal pain hindering adequate gastric ultrasound
* patients with a Percutaneous Endoscopic Gastrostomy catheter

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients are selected from a surgical ward, patients recover from liver surgery, colorectal or hyperthermic intraperitoneal chemotherapy (HIPEC) surgery, pancreatic surgery, or other gastro-intestinal abdominal procedures
Sampling Method: Non-Probability Sample
Enrollment: 135 (Estimated)
Dates: Start 2024-04-22 (Actual); Primary Completion 2024-11-16 (Estimated); Study Completion 2024-12-24 (Estimated)

PRIMARY OUTCOMES:
Feasibility of gastric ultrasound in terms of practicality | through study completion, for 6 months
  Practicality of gastric ultrasound will be measured by the length in minutes.
Feasibility of gastric ultrasound in terms of usability | through study completion, for 6 months
  The Dutch-System Usability Scale will be used to assess usability
Feasibility of gastric ultrasound in terms of acceptability perceived by patients | through study completion, for 6 months
  Acceptability will be measured by the patients' perspective towards undergoing gastric ultrasound during recovery after surgery.
Feasibility of gastric ultrasound in terms of demand | through study completion, for 6 months
  Demand will be measured by indications for gastric ultrasound and the change for successful image acquisition. Indications involve a description of clinical signs that were present during the gastric ultrasound performance. Each attempt for gastric ultrasound will be counted, afterwards adequate images will be counted. Change for succesfull image acquisition wil be calculated by adequate images divided by numbers of attemps. Both values indicate the demand according to its definition
Feasibility of Gastric ultrasound in terms of nurses accuracy and nurses confidence | through study completion, an average of 6 months
  The nurses accuracy and nurses' confidence to perform gastric ultrasound will be assessed. Accuracy will be measured by validating the ultrasound findings independently by expert sonographers and the nurses for their peers, determining inter-rater reliability.
Feasibility of gastric ultrasound in terms of acceptability perceived by nurses | through study completion, for 6 months
  Acceptability will be measured by the nurses' perspective towards the acceptability of gastric ultrasound. This is measured with the Theoretical Framework of Acceptability-based (TFA) questionnaire which is modified to assess the acceptability of gastric ultrasound during recovery after surgery.

CONTACTS AND LOCATIONS:
Overall Officials: Harm HJ van Noort, PhD, Principal Investigator — Radboud University Medical Center
Locations (2):
- Netherlands (2):
  - RadboudUMC, Nijmegen, Gelderland
  - Radboudumc, Nijmegen

IPD SHARING:
Plan to Share IPD: Undecided
Data will be stored according to hospital guidelines and shared upon reasonable request

REFERENCES:
- [Background] Van de Putte P, Perlas A. Ultrasound assessment of gastric content and volume. Br J Anaesth. 2014 Jul;113(1):12-22. doi: 10.1093/bja/aeu151. Epub 2014 Jun 3. PMID 24893784
- [Background] Lamm R, Collins M, Bloom J, Joel M, Iosif L, Park D, Reny J, Schultz S, Yeo CJ, Beausang D, Schwenk ES, Costanzo C, Phillips BR. Postoperative Handheld Gastric Point-of-Care Ultrasound and Delayed Bowel Function. J Am Coll Surg. 2023 Apr 1;236(4):554-559. doi: 10.1097/XCS.0000000000000536. Epub 2023 Jan 5. PMID 36602237
- [Background] Lamm R, Bloom J, Collins M, Goldman D, Beausang D, Costanzo C, Schwenk ES, Phillips B. A Role for Gastric Point of Care Ultrasound in Postoperative Delayed Gastrointestinal Functioning. J Surg Res. 2022 Aug;276:92-99. doi: 10.1016/j.jss.2022.02.028. Epub 2022 Mar 24. PMID 35339785
- [Background] Brotfain E, Erblat A, Luft P, Elir A, Gruenbaum BF, Livshiz-Riven I, Koyfman A, Fridrich D, Koyfman L, Friger M, Grivnev A, Zlotnik A, Klein M. Nurse-performed ultrasound assessment of gastric residual volume and enteral nasogastric tube placement in the general intensive care unit. Intensive Crit Care Nurs. 2022 Apr;69:103183. doi: 10.1016/j.iccn.2021.103183. Epub 2021 Dec 16. PMID 34924254
- [Background] Arzola C, Carvalho JC, Cubillos J, Ye XY, Perlas A. Anesthesiologists' learning curves for bedside qualitative ultrasound assessment of gastric content: a cohort study. Can J Anaesth. 2013 Aug;60(8):771-9. doi: 10.1007/s12630-013-9974-y. Epub 2013 May 24. PMID 23703533
- [Background] Cozza V, Barberis L, Altieri G, Donatelli M, Sganga G, La Greca A. Prediction of postoperative nausea and vomiting by point-of-care gastric ultrasound: can we improve complications and length of stay in emergency surgery? A cohort study. BMC Anesthesiol. 2021 Aug 31;21(1):211. doi: 10.1186/s12871-021-01428-0. PMID 34465303